CLINICAL TRIAL: NCT01568866
Title: A Randomized, Open-label, Phase 3 Study of Carfilzomib Plus Dexamethasone vs. Bortezomib Plus Dexamethasone in Patients With Relapsed Multiple Myeloma
Brief Title: Phase 3 Study With Carfilzomib and Dexamethasone Versus Bortezomib and Dexamethasone for Relapsed Multiple Myeloma Patients
Acronym: ENDEAVOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-003; 2012-000128-16 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; relapsed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carfilzomib plus Dexamethasone (Experimental): Participants received 20 mg/m² carfilzomib administered by intravenous (IV) infusion on Days 1 and 2 of Cycle 1, followed by 56 mg/m² on Days 8, 9, 15, and 16 of Cycle 1 and for each 28-day cycle thereafter. Additionally, participants received 20 mg dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28 day cycle.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone
- Bortezomib plus Dexamethasone (Active Comparator): Participants received bortezomib 1.3 mg/m² administered IV or subcutaneously (SC) on Days 1, 4, 8, and 11 of a 21-day cycle plus dexamethasone 20 mg administered on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib is administered over 30 minutes as an infusion.
  Other Names: PR-171; Krypolis
  Arms: Carfilzomib plus Dexamethasone
Drug: Bortezomib — Bortezomib is administered as a 3-5 second bolus IV injection or SC injection (in accordance with regulatory approval)
  Other Names: Velcade
  Arms: Bortezomib plus Dexamethasone
Drug: Dexamethasone — Tablet for oral administration; On days when carfilzomib or bortezomib was administered, the dexamethasone was to be given 30 minutes to 4 hours prior to the carfilzomib or bortezomib dose.

SUMMARY:
The primary objective of this study was to compare progression-free survival in patients with multiple myeloma who relapsed after 1 to 3 prior therapies treated with carfilzomib plus dexamethasone or bortezomib plus dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma with relapsing or progressing disease at study entry.
2. Patients must have evaluable multiple myeloma with, at least one of the following (assessed within 21 days prior to randomization):

   * Serum M-protein ≥ 0.5 g/dL, or
   * Urine M-protein ≥ 200 mg/24 hour, or
   * In patients without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal serum kappa/lamda ratio, or
   * For immunoglobulin (Ig) A patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA) ≥ 750 mg/dL (0.75 g/dL).
3. Patients must have documented at least partial response (PR) to at least 1 line of prior therapy. PR documentation can be based on Investigator assessment.
4. Received 1, but no more than 3 prior treatment regimens or lines of therapy for multiple myeloma. (Induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as one line of therapy).
5. Prior therapy with Velcade is allowed as long as the patient had at least a PR to prior Velcade therapy, was not removed from Velcade therapy due to toxicity, and will have at least a 6 month Velcade treatment-free interval from last dose received until first study treatment. (Patients may receive maintenance therapy with drugs that are not in the proteasome inhibitor class during this 6 month Velcade treatment-free interval).
6. Prior therapy with carfilzomib is allowed as long as the patient had at least a PR to prior carfilzomib therapy, was not removed from carfilzomib therapy due to toxicity, and had at least a 6-month carfilzomib treatment-free interval from last dose received until first study treatment. (Patients may receive maintenance therapy with drugs that are not in the proteasome inhibitor class during this 6 month carfilzomib treatment-free interval). The exception to this is patients randomized or previously randomized in any other Onyx-Sponsored Phase 3 trial.
7. Males and females ≥ 18 years of age.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
9. Adequate hepatic function within 21 days prior to randomization, with bilirubin < 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN.
10. Left ventricular ejection fraction (LVEF) ≥ 40%.
11. Absolute neutrophil count (ANC) ≥ 1000/mm³ within 21 days prior to randomization. Screening ANC should be independent of growth factor support for ≥ 1 week.
12. Hemoglobin ≥ 8.0 g/dL within 21 days prior to randomization. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed, however most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin.
13. Platelet count ≥ 50,000/mm³ (≥ 30,000/mm³ if myeloma involvement in the bone marrow is > 50%) within 21 days prior to randomization. Patients should not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count.
14. Calculated or measured creatinine clearance (CrCl) of ≥ 15 mL/min within 21 days prior to randomization. Calculation should be based on standard formula such as the Cockcroft and Gault:

    [(140 - Age) x Mass (kg) / (72 x Creatinine mg/dL)]; multiply result by 0.85 if female.
15. Written informed consent in accordance with federal, local, and institutional guidelines.
16. Female patients of child-bearing potential (FCBP) must have a negative serum pregnancy test within 21 days prior to randomization and agree to use an effective method of contraception during and for 3 months following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations). FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
17. Male patients must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a FCBP.

Exclusion Criteria:

1. Multiple Myeloma of IgM subtype.
2. Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 14 days prior to randomization.
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
4. Plasma cell leukemia or circulating plasma cells ≥ 2 × 10^9/L.
5. Waldenstrom's Macroglobulinemia.
6. Patients with known amyloidosis.
7. Chemotherapy with approved or investigational anticancer therapeutics within 21 days prior to randomization.
8. Patients randomized or previously randomized in any other Onyx-Sponsored Phase 3 trial.
9. Focal radiation therapy within 7 days prior to randomization. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to randomization (i.e., prior radiation must have been to less than 30% of the bone marrow).
10. Immunotherapy within 21 days prior to randomization.
11. Major surgery (excluding kyphoplasty) within 28 days prior to randomization.
12. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within four months prior to randomization.
13. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents within 14 days prior to randomization.
14. Known human immunodeficiency (HIV) seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen [SAg] or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed).
15. Patients with known cirrhosis.
16. Second malignancy within the past 3 years except:

    * adequately treated basal cell or squamous cell skin cancer
    * carcinoma in situ of the cervix
    * prostate cancer < Gleason score 6 with stable prostate-specific antigen (PSA) over 12 months
    * breast carcinoma in situ with full surgical resection
    * treated medullary or papillary thyroid cancer
17. Patients with myelodysplastic syndrome.
18. Significant neuropathy (Grades 3 to 4, or Grade 2 with pain) within 14 days prior to randomization.
19. Female patients who are pregnant or lactating.
20. Known history of allergy to Captisol(a cyclodextrin derivative used to solubilize carfilzomib).
21. Patients with hypersensitivity to carfilzomib, Velcade, boron, or mannitol.
22. Patients with contraindication to dexamethasone.
23. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
24. Ongoing graft-vs-host disease.
25. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2014-11-10 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (241):
- United States (27):
  - Providence St. Joseph Medical Center, Burbank, California
  - UCSD Moore Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Central Coast Medical Oncology Group, Santa Maria, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - MAB Oncology/Hematology, Melbourne, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Hematology Oncology of Indiana, PC, Indianapolis, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Associates in Oncology/Hematology PC, Rockville, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Kansas, Kansas City, Missouri
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Clinical Research Alliance Inc., New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Section on Hematology and Oncology, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hematology/Oncology Associates of SC, Greenville, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - The Methodist Cancer Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Australia (21):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Saint George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Haematology & Oncology Clinics of Australia, South Brisbane, Queensland
  - Haematology and Oncology Clinics of Australia at Chermside, South Brisbane, Queensland
  - Haematology and Oncology Clinics of Australia at Wesley, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Saint Vincent's Hospital, East Melbourne, Victoria
  - Western Hospital, Footscray, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Krankenhaus der Elisabethinen Linz, I Interne Abteilung, Linz, Upper Austria
  - Wilhelminenspital der Stadt Wien, Vienna, Vienna
- Belgium (6):
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir, Namur
  - Universitair Ziekenhuis Gent, Ghent, Oost-vlaanderen
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
- Brazil (9):
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Clínica de Oncologia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hemocentro Campinas-Unicamp, Campinas, São Paulo
  - Hospital Universitário Clementino Fraga Filho da Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Instituto Centros Oncológicos Integrados de Educação e Pesquisa, Rio de Janeiro
  - Instituto Nacional do Câncer-INCA, Rio de Janeiro
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo
- Bulgaria (4):
  - Military Medical Academy Hospital for Active Treatment, Sofia, Sofia
  - Shato, Ead, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment, "Sveta Marina'', Varna
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (6):
  - Fakultní nemocnice Královské Vinohrady, Prague, Prague
  - Fakultní nemocnice Olomouc, Olomouc, Severomoravsky KRAJ
  - FN Ostrava, Ostrava, Severomoravsky KRAJ
  - Fakultní nemocnice Hradec Králové, Hradec Kralové, Vychodocesky KRAJ
  - Fakultní nemocnice Brno, Brno
  - Všeobecná fakultní nemocnice v Praze, Prague
- France (12):
  - Centre Hospitalier de la Cote Basque, Bayonne, Aquitaine
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Brest, Brest, Brittany Region
  - Centre Hospitalier Universitaire de Rennes, Hôpital Pontchaillou, Rennes, Brittany Region
  - Hopital Hotel-Dieu - Service d'Hematologie, Nantes, Cedex 1
  - Centre Henri-Becquerel, Rouen, Haute-normandie
  - Hôpital Claude Huriez, Lille, Hauts-de-France
  - Hôpital Hôtel-Dieu, Nantes, Pays de la Loire Region
  - Institut Paoli Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de Versailles, Le Chesnay, Île-de-France Region
  - Hôpital Saint Louis, Paris, Île-de-France Region
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
- Germany (15):
  - Universitätsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Medizinische Klinik der Universität Würzburg, Würzburg, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg / Saar, Saarland
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinikum Carl Gustav Carus, Med. Klinik und Poliklinik I, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Alexandra General Hospital, Athens, Attica, Greece
- Hungary (7):
  - Pécsi Tudományegyetem, Pécs, Baranya
  - Bács-Kiskun Megyei Kórház Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, Kecskemét, Bács-Kiskun county
  - Szegedi Tudományegyetem, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Egyesített Szent István és Szent László Kórház-Rendelointézet, Budapest
  - Somogy Megyei Kaposi Mac okato Korhoz, Kaposvár
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Israel (5):
  - Rambam Health Corp., Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center at Tel Hashomer, Tel Litwinsky
- Italy (14):
  - IRCCS Centro di Riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture, Potenza
  - Azienda Ospedaliero-Univesitaria San Luigi Gonzaga, Orbassano, Torino
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Novara
  - Azienda Unità Sanitaria Locale di Piacenza-Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Ospedaliera Pisana Ospedale Santa Chiara, Pisa
  - Aienda Policknico Umberto I di Roma, Roma
  - Azienda Policknico Umberto l di Roma, Roma
  - Università Tor Vergata Ospedale Sant Eugenio, Roma
  - Azienda Ospedaliera Universitaria Senese - Policlinico S. Maria alle Scotte, Siena
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (24):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Nishigunma National Hospital, Shibukawa, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of Japanese Foundation For Cancer Research, Koto-ku, Tokyo
  - Toranornon Hospital, Shinagawa, Tokyo
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Social Insurance Kyoto Hospital of All Japan Federation of Social Insurance Associations, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Tokushima Prefectural Central Hospital, Tokushima
  - Japanese Red Cross Medical Center, Tokyo
- New Zealand (5):
  - North Shore Hospital, North Shore, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - Auckland City Hospital, Grafton, Aukland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Poland (7):
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im K. Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - Specjalistyczny Szpital Miejski im. Mikolaja Kopernika, Torun, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Zamojski Szpital Niepubliczny Sp. z o.o., Zamość, Lublin Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespól Szpitali Miejskich, Chorzów, Silesian Voivodeship
- Romania (5):
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest, București
  - Policlinica de Diagnostic Rapid SA, Compartiment Medical Oncologie-Hematologie, Brasov
  - Spitalul Clinic Judetean de Urgenta Brasov (Bumbea, Horia), Brasov
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Regional de Oncologie Iasi, Iași
- Russia (9):
  - Republican Clinical Hospital #1, Izhevsk
  - City Clinical Hospital n.a. S. P. Botkin, Moscow
  - Non-state Healthcare Institution "N.A. Semashko Central Clinical Hospital #2 of JSC "Russian Railway, Moscow
  - Ryazan Regional Clinical Hospital, Ryazan
  - Clinical Hospital Number 31, Saint Petersburg
  - Federal Almazov Medical Research Centre, Saint Petersburg
  - FGU Russian Scientific Research Institute of Hematology and Transfusiology, Saint Petersburg
  - First Saint Petersburg I.P. Pavlov State Medical University, Saint Petersburg
  - GUZ Samara Regional Clinical Hospital n.a. M.I. Kalinin, Samara
- Singapore (3):
  - National University Cancer Institute, Singapore
  - Singapore General Hospital, Singapore
  - Singapore Oncology Consultants, Singapore
- Univerzitná nemocnica Bratislava, Bratislava, Slovakia
- South Korea (9):
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Pusan, Gyeongsangnam-do
  - Kyungpook National University Hospital, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (10):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Institut Universitari Dexeus, Barcelona
  - Centro Integral Oncológico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fé de Valencia, Valencia
- Taiwan (6):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-LinKou Branch, Taoyuan District
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok, Bangkok Metropolis
  - Ramathibodi Hospital, Bangkok, Bangkok Metropolis
  - Srinagarind Hospital, Khon Kaen
- Ukraine (12):
  - City Hematology Center, Dnipro, Dnipropretrovsk
  - Municipal Institution of Health Protection "Clinical Hospital #8", Kharkiv, Kharkivs’ka Oblast’
  - Cherkassy Regional Oncology Center, Cherkassy
  - MI "Dnipropetrovsk City Multifield Clinical Hospital #4" of Dnipropetrovsk Regional Council", City Hematology Center, Dnipropetrovsk
  - Institute of Urgent and Reparative Surgury of Ukraine Academy of Medical Sciences, Donetsk
  - Khmelnytsky Regional Clinical Hospital, Khmelnytsky
  - Khmelnytsky Regional Hospital, Department of Hematology, Khmelnytsky
  - National Institute of Cancer, Oncohematology Department, Kiev
  - Kyiv Bone Marrow Transplantation Center, Kyiv
  - Lviv Regional Oncology Dispensary, Lviv
  - Lviv State Oncology Regional Treatment-Prophylactic Center, Department of Chemotherapy, Lviv
  - Regional Clinical Hospital, Mykolayiv
- United Kingdom (9):
  - Royal Free Hospital, London, England
  - University College Hospital, London, England
  - Manchester Royal Infirmary, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Royal Marsden Hospital, Surrey, England
  - Royal Wolverhampton Hospitals Trust, Wolverhampton, England

REFERENCES:
- [Background] Moreau P, Joshua D, Chng WJ, Palumbo A, Goldschmidt H, Hajek R, Facon T, Ludwig H, Pour L, Niesvizky R, Oriol A, Rosinol L, Suvorov A, Gaidano G, Pika T, Weisel K, Goranova-Marinova V, Gillenwater HH, Mohamed N, Aggarwal S, Feng S, Dimopoulos MA. Impact of prior treatment on patients with relapsed multiple myeloma treated with carfilzomib and dexamethasone vs bortezomib and dexamethasone in the phase 3 ENDEAVOR study. Leukemia. 2017 Jan;31(1):115-122. doi: 10.1038/leu.2016.186. Epub 2016 Jul 4. PMID 27491641
- [Background] Chng WJ, Goldschmidt H, Dimopoulos MA, Moreau P, Joshua D, Palumbo A, Facon T, Ludwig H, Pour L, Niesvizky R, Oriol A, Rosinol L, Suvorov A, Gaidano G, Pika T, Weisel K, Goranova-Marinova V, Gillenwater HH, Mohamed N, Feng S, Aggarwal S, Hajek R. Carfilzomib-dexamethasone vs bortezomib-dexamethasone in relapsed or refractory multiple myeloma by cytogenetic risk in the phase 3 study ENDEAVOR. Leukemia. 2017 Jun;31(6):1368-1374. doi: 10.1038/leu.2016.390. Epub 2016 Dec 27. PMID 28025582
- [Background] Dimopoulos MA, Goldschmidt H, Niesvizky R, Joshua D, Chng WJ, Oriol A, Orlowski RZ, Ludwig H, Facon T, Hajek R, Weisel K, Hungria V, Minuk L, Feng S, Zahlten-Kumeli A, Kimball AS, Moreau P. Carfilzomib or bortezomib in relapsed or refractory multiple myeloma (ENDEAVOR): an interim overall survival analysis of an open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1327-1337. doi: 10.1016/S1470-2045(17)30578-8. Epub 2017 Aug 23. PMID 28843768
- [Background] Ludwig H, Dimopoulos MA, Moreau P, Chng WJ, Goldschmidt H, Hajek R, Facon T, Pour L, Niesvizky R, Oriol A, Rosinol L, Suvorov A, Gaidano G, Pika T, Weisel K, Goranova-Marinova V, Palumbo A, Gillenwater HH, Mohamed N, Aggarwal S, Feng S, Joshua D. Carfilzomib and dexamethasone vs bortezomib and dexamethasone in patients with relapsed multiple myeloma: results of the phase 3 study ENDEAVOR (NCT01568866) according to age subgroup. Leuk Lymphoma. 2017 Oct;58(10):2501-2504. doi: 10.1080/10428194.2017.1298755. Epub 2017 Mar 17. No abstract available. PMID 28306371
- [Background] Chari A, Stewart AK, Russell SD, Moreau P, Herrmann J, Banchs J, Hajek R, Groarke J, Lyon AR, Batty GN, Ro S, Huang M, Iskander KS, Lenihan D. Analysis of carfilzomib cardiovascular safety profile across relapsed and/or refractory multiple myeloma clinical trials. Blood Adv. 2018 Jul 10;2(13):1633-1644. doi: 10.1182/bloodadvances.2017015545. PMID 29991494
- [Background] Dimopoulos M, Siegel D, White DJ, Boccia R, Iskander KS, Yang Z, Kimball AS, Mezzi K, Ludwig H, Niesvizky R. Carfilzomib vs bortezomib in patients with multiple myeloma and renal failure: a subgroup analysis of ENDEAVOR. Blood. 2019 Jan 10;133(2):147-155. doi: 10.1182/blood-2018-06-860015. Epub 2018 Nov 26. PMID 30478094
- [Background] Facon T, Niesvizky R, Mateos MV, Siegel D, Rosenbaum C, Bringhen S, Weisel K, Ho PJ, Ludwig H, Kumar S, Wang K, Obreja M, Yang Z, Klippel Z, Mezzi K, Goldrick A, Tekle C, Dimopoulos MA. Efficacy and safety of carfilzomib-based regimens in frail patients with relapsed and/or refractory multiple myeloma. Blood Adv. 2020 Nov 10;4(21):5449-5459. doi: 10.1182/bloodadvances.2020001965. PMID 33166401
- [Background] Hari P, Mateos MV, Abonour R, Knop S, Bensinger W, Ludwig H, Song K, Hajek R, Moreau P, Siegel DS, Feng S, Obreja M, Aggarwal SK, Iskander K, Goldschmidt H. Efficacy and safety of carfilzomib regimens in multiple myeloma patients relapsing after autologous stem cell transplant: ASPIRE and ENDEAVOR outcomes. Leukemia. 2017 Dec;31(12):2630-2641. doi: 10.1038/leu.2017.122. Epub 2017 Apr 25. PMID 28439109
- [Background] Leleu X, Martin TG, Einsele H, Lyons RM, Durie BGM, Iskander KS, Ailawadhi S. Role of Proteasome Inhibitors in Relapsed and/or Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2019 Jan;19(1):9-22. doi: 10.1016/j.clml.2018.08.016. Epub 2018 Sep 5. PMID 30287200
- [Background] Ludwig H, Moreau P, Dimopoulos MA, Mateos MV, Kaiser M, Hajek R, Feng S, Cocks K, Buchanan J, Weisel K. Health-related quality of life in the ENDEAVOR study: carfilzomib-dexamethasone vs bortezomib-dexamethasone in relapsed/refractory multiple myeloma. Blood Cancer J. 2019 Feb 22;9(3):23. doi: 10.1038/s41408-019-0181-0. PMID 30796199
- [Background] Mateos MV, Goldschmidt H, San-Miguel J, Mikhael J, DeCosta L, Zhou L, Obreja M, Blaedel J, Szabo Z, Leleu X. Carfilzomib in relapsed or refractory multiple myeloma patients with early or late relapse following prior therapy: A subgroup analysis of the randomized phase 3 ASPIRE and ENDEAVOR trials. Hematol Oncol. 2018 Apr;36(2):463-470. doi: 10.1002/hon.2499. Epub 2018 Feb 15. PMID 29446103
- [Background] Moreau P, Stewart KA, Dimopoulos M, Siegel D, Facon T, Berenson J, Raje N, Berdeja JG, Orlowski RZ, Yang H, Ma H, Klippel Z, Zahlten-Kumeli A, Mezzi K, Iskander K, Mateos MV. Once-weekly (70 mg/m2 ) vs twice-weekly (56 mg/m2 ) dosing of carfilzomib in patients with relapsed or refractory multiple myeloma: A post hoc analysis of the ENDEAVOR, A.R.R.O.W., and CHAMPION-1 trials. Cancer Med. 2020 May;9(9):2989-2996. doi: 10.1002/cam4.2945. Epub 2020 Feb 28. PMID 32108443
- [Background] Dimopoulos MA, Moreau P, Iida S, Huang SY, Takezako N, Chng WJ, Zahlten-Kumeli A, Sersch MA, Li J, Huang M, Lee JH. Outcomes for Asian patients with multiple myeloma receiving once- or twice-weekly carfilzomib-based therapy: a subgroup analysis of the randomized phase 3 ENDEAVOR and A.R.R.O.W. Trials. Int J Hematol. 2019 Oct;110(4):466-473. doi: 10.1007/s12185-019-02704-z. Epub 2019 Aug 6. PMID 31388932
- [Background] Goldschmidt H, Moreau P, Ludwig H, Niesvizky R, Chng WJ, Joshua D, Weisel K, Spencer A, Orlowski RZ, Feng S, Iskander KS, Dimopoulos MA. Carfilzomib-dexamethasone versus subcutaneous or intravenous bortezomib in relapsed or refractory multiple myeloma: secondary analysis of the phase 3 ENDEAVOR study. Leuk Lymphoma. 2018 Jun;59(6):1364-1374. doi: 10.1080/10428194.2017.1376743. Epub 2017 Sep 22. PMID 28937327
- [Background] Jakubowiak AJ, Houisse I, Majer I, Benedict A, Campioni M, Panjabi S, Ailawadhi S. Cost-effectiveness of carfilzomib plus dexamethasone compared with bortezomib plus dexamethasone for patients with relapsed or refractory multiple myeloma in the United States. Expert Rev Hematol. 2017 Dec;10(12):1107-1119. doi: 10.1080/17474086.2017.1391088. PMID 29027825
- [Background] Weisel K, Mateos MV, Gay F, Delforge M, Cook G, Szabo Z, Desgraz R, DeCosta L, Moreau P. Efficacy and safety profile of deep responders to carfilzomib-based therapy: a subgroup analysis from ASPIRE and ENDEAVOR. Leukemia. 2021 Jun;35(6):1732-1744. doi: 10.1038/s41375-020-01049-5. Epub 2020 Oct 16. PMID 33067574
- [Background] Weisel K, Majer I, DeCosta L, Oriol A, Goldschmidt H, Ludwig H, Campioni M, Szabo Z, Dimopoulos M. Carfilzomib and dexamethasone versus eight cycles of bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma: an indirect comparison using data from the phase 3 ENDEAVOR and CASTOR trials. Leuk Lymphoma. 2020 Jan;61(1):37-46. doi: 10.1080/10428194.2019.1648806. Epub 2019 Oct 22. PMID 31640435
- [Background] Orlowski RZ, Moreau P, Niesvizky R, Ludwig H, Oriol A, Chng WJ, Goldschmidt H, Yang Z, Kimball AS, Dimopoulos M. Carfilzomib-Dexamethasone Versus Bortezomib-Dexamethasone in Relapsed or Refractory Multiple Myeloma: Updated Overall Survival, Safety, and Subgroups. Clin Lymphoma Myeloma Leuk. 2019 Aug;19(8):522-530.e1. doi: 10.1016/j.clml.2019.04.018. Epub 2019 May 2. PMID 31160237
- [Derived] Majer IM, Castaigne JG, Palmer S, DeCosta L, Campioni M. Modeling Covariate-Adjusted Survival for Economic Evaluations in Oncology. Pharmacoeconomics. 2019 May;37(5):727-737. doi: 10.1007/s40273-018-0759-6. PMID 30610657
- [Derived] Rosenthal A, Luthi J, Belohlavek M, Kortum KM, Mookadam F, Mayo A, Fonseca R, Bergsagel PL, Reeder CB, Mikhael JR, Stewart AK. Carfilzomib and the cardiorenal system in myeloma: an endothelial effect? Blood Cancer J. 2016 Jan 15;6(1):e384. doi: 10.1038/bcj.2015.112. PMID 26771810
- [Derived] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with relapsed multiple myeloma were enrolled between 20 June 2012 and 30 June 2014 at 198 centers in 27 countries in Europe, North America, South America, and the Asia-Pacific region.
  Results are reported as of the data cut-off date of 03 January 2017, the pre-specified 2nd interim analysis of the secondary endpoint of overall survival.
Pre-assignment Details: Randomization was stratified by previous proteasome inhibitor therapy (yes vs no), previous lines of treatment (1 vs 2 or 3), International Staging System stage (I vs II-III), and planned route of bortezomib administration (intravenous vs subcutaneous) if randomly assigned to the bortezomib group.
Groups:
- Bortezomib + DEX: Participants received bortezomib 1.3 mg/m² administered intravenously (IV) or subcutaneously (SC) on Days 1, 4, 8, and 11 of a 21-day cycle plus dexamethasone (DEX) 20 mg administered on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle.
- Carfilzomib + DEX: Participants received 20 mg/m² carfilzomib administered by IV infusion on Days 1 and 2 of Cycle 1, followed by 56 mg/m² on Days 8, 9, 15, and 16 of Cycle 1 and for each 28-day cycle thereafter. Additionally, participants received 20 mg dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28 day cycle.
Period: Overall Study
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Started | 465 | 464
Received Treatment | 456 | 463
Completed | 27 (Indicates participants still receiving treatment) | 48 (Indicates participants still receiving treatment)
Not Completed | 438 | 416
Not completed — Disease Progression | 208 | 183
Not completed — Adverse Event | 94 | 96
Not completed — Patient Request | 55 | 71
Not completed — Physician Decision | 40 | 32
Not completed — Withdrawal by Subject | 19 | 11
Not completed — Death | 10 | 18
Not completed — Protocol Non-compliance | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Randomized but Not Dosed | 9 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (all randomized participants)
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX | Total
Number analyzed (Participants) | 465 | 464 | 929
Age, Continuous [Median (Full Range); unit: years] | 65.0 [30.0 to 88.0] | 65.0 [35.0 to 89.0] | 65.0 [30.0 to 89.0]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 210 | 223 | 433
  65 -74 years | 189 | 164 | 353
  ≥ 75 years | 66 | 77 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 224 | 460
  Male | 229 | 240 | 469
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 353 | 348 | 701
  Black | 9 | 8 | 17
  Asian | 57 | 56 | 113
  Native Hawaiian/Other Pacific Islander | 0 | 2 | 2
  Not Reported | 45 | 50 | 95
  Multiple | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 232 | 221 | 453
    1 (Restrictive but ambulatory) | 203 | 211 | 414
    2 (Ambulatory but unable to work) | 30 | 32 | 62
Stratification Factor: Prior Proteasome Inhibitor Treatment [Count of Participants; unit: Participants]
  Carfilzomib or bortezomib | 253 | 252 | 505
  No prior carfilzomib or bortezomib | 212 | 212 | 424
Stratification Factor: Lines of Prior Treatment [Count of Participants; unit: Participants]
  1 line | 229 | 231 | 460
  2 or 3 lines | 236 | 233 | 469
Stratification Factor: International Staging System (ISS) Stage [Count of Participants; unit: Participants] — The International Staging System (ISS) for myeloma was published by the International Myeloma Working Group:
  * Stage I: β2-microglobulin (β2M) < 3.5 mg/L, albumin >= 3.5 g/dL
  * Stage II: β2M < 3.5 mg/L and albumin < 3.5 g/dL; or β2M 3.5 mg/L - 5.5 mg/L irrespective of the serum albumin
  * Stage III: β2M ≥ 5.5 mg/L
  Participants
    Stage I | 204 | 205 | 409
    Stage II or III | 261 | 259 | 520
Stratification Factor: Route of Bortezomib Administration [Count of Participants; unit: Participants] — The route of bortezomib administration (IV versus SC) was made in accordance with local regulatory approved route of administration. The value for this variable was selected for all participants prior to randomization to treatment group in order to balance the baseline characteristics that led to the choice of the particular route of bortezomib administration between the 2 arms.
  Participants
    Intravenous | 108 | 108 | 216
    Subcutaneous | 357 | 356 | 713

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from randomization to the earlier of disease progression or death due to any cause. Participants were evaluated for disease response and progression according to the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC) as assessed by an Independent Review Committee (IRC).
  Median PFS was estimated using the Kaplan-Meier method. Participants with no baseline disease assessments, starting a new anticancer therapy before documentation of disease progression or death, death or disease progression immediately after more than 1 consecutively missed disease assessment visit, or alive without documentation of disease progression before the data cut-off date were censored.
Time Frame: From randomization until the data cut-off date of 10 November 2014; median follow-up time for PFS was 11.1.and 11.9 months in the bortezomib and carfilzomib arms respectively
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 465 | 464
months | 9.4 [8.4 to 10.4] | 18.7 [15.6 to NA] — Could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: Bortezomib + DEX vs Carfilzomib + DEX; The PFS interim analysis was to be performed using a group sequential monitoring plan. The monitoring plan included an O'Brien-Fleming type of efficacy stopping boundary constructed using the Lan-DeMets alpha spending function to ensure a 1-sided Type I error rate ≤ 0.025; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank; Log rank test stratified by the randomization stratification factors; Hazard Ratio (HR) = 0.533, 95% CI 2-sided [0.437 to 0.651] — The hazard ratio (carfilzomib/bortezomib) was estimated using a Cox proportional hazards model stratified by prior proteasome inhibitor treatment, lines of prior treatment, ISS stage, and choice of route of bortezomib administration

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to the date of death (whatever the cause). Participants who were alive or lost to follow-up as of the data analysis cut-off date were censored at the patient's date of last contact (last known to be alive).
  Median overall survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization until the data cut-off date of 03 January 2017; median follow-up time for OS was 36.9 and 37.5 months for each treatment group respectively.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 465 | 464
months | 40.0 [32.6 to 42.3] | 47.6 [42.5 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Bortezomib + DEX vs Carfilzomib + DEX; The second interim analysis of overall survival was to be conducted after 394 events had been reached. A one-sided significance level was determined using the O'Brien-Fleming-type α spending function based on the actual number of events (α=0.0123); Test type: Superiority or Other; p = 0.0100, Stratified Log Rank — The multiplicity in testing secondary endpoints was adjusted per group using the sequential Holm procedure to preserve the family-wise error rate at 0.025; Log rank test stratified by the randomization stratification factors; Hazard Ratio (HR) = 0.791, 95% CI 2-sided [0.648 to 0.964] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response
Description: Disease response was evaluated according to the IMWG-URC by the IRC. Overall response was defined as the percentage of participants with a best overall response of partial response (PR), very good PR (VGPR), complete response (CR) or stringent CR (sCR).
  sCR: As for CR, normal serum free light chain (SFLC) ratio and no clonal cells in bone marrow (BM).
  CR: No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in BM biopsy; VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-protein with urine M-protein <100 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
  PR: ≥ 50% reduction of serum M-protein and reduction in urine M-protein by ≥ 90% or to < 200 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
Time Frame: Disease response was assessed every 28 days until end of treatment or the data cut-off date of 10 November 2014; median duration of treatment was 27 weeks in the bortezomib group and 40 weeks in the carfilzomib treatment group.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 465 | 464
percentage of participants | 62.6 [58.0 to 67.0] | 76.9 [72.8 to 80.7]
Statistical Analysis 1: Comparison: Bortezomib + DEX vs Carfilzomib + DEX; Test type: Superiority or Other; p < 0.0001, Stratified Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Cochran-Mantel-Haenszel test stratified by the randomization stratification factors; Odds Ratio (OR) = 2.032, 95% CI 2-sided [1.519 to 2.718] — The odds ratio (carfilzomib/bortezomib) was calculated using the Cochran-Mantel-Haenszel method stratified by prior proteasome inhibitor treatment, lines of prior treatment, ISS stage, and choice of route of bortezomib administration

4. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was calculated for participants who achieved an sCR, CR, VGPR, or PR. Duration of response is defined as the time from first evidence of PR or better to confirmation of disease progression or death due to any cause. Median duration of response was estimated using the Kaplan-Meier method. Participants with no baseline disease assessments, starting a new anticancer therapy before documentation of disease progression or death, death or disease progression immediately after more than 1 consecutively missed disease assessment visit, or alive without documentation of disease progression before the data cut-off date were censored.
Time Frame: From randomization until the data cut-off date of 10 November 2014; median follow-up time for DOR was 9.4 and 10.4 months for each treatment group respectively.
Population: Intent-to-treat population with an overall response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 291 | 357
months | 10.4 [9.3 to 13.8] | 21.3 [21.3 to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Percentage of Participants With ≥ Grade 2 Peripheral Neuropathy
Description: Neuropathy events were defined as Grade 2 or higher peripheral neuropathy as specified by peripheral neuropathy Standardised Medical Dictionary for Regulatory Activities (MedDRA) Query, narrow (scope) (SMQN) terms.
  Peripheral neuropathy was assessed by neurologic exam and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03:
  Grade 1: Asymptomatic; Grade 2: Moderate symptoms, limiting instrumental activities of daily living (ADL) Grade 3: Severe symptoms; limiting self-care ADL; Grade 4: Life-threatening consequences, urgent intervention indicated; Grade 5: Death.
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug as of the data cut-off date of 10 November 2014; median duration of treatment was 27 weeks in the bortezomib group and 40 weeks in the carfilzomib treatment group.
Population: Safety population (all participants who received at least 1 dose of study treatment)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 456 | 463
percentage of participants | 32.0 [27.7 to 36.3] | 6.0 [3.9 to 8.2]
Statistical Analysis 1: Comparison: Bortezomib + DEX vs Carfilzomib + DEX; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.137, 95% CI 2-sided [0.089 to 0.210] — The odds ratio (carfilzomib/bortezomib) was estimated using the unconditional Cochran-Mantel-Haenszel method

6. Secondary Outcome: Percentage of Participants With a Significant Reduction in Left Ventricular Ejection Fraction (LVEF)
Description: A significant reduction in LVEF was defined as a ≥ 10% decrease (absolute change) from baseline in participants whose baseline LVEF is ≤ 55%.
  For participants with LVEF > 55% at baseline, a significant change was defined as a decrease in LVEF to < 45%.
Time Frame: Baseline and 24 weeks
Population: Cardiopulmonary Safety Evaluable subgroup (all randomized participants who enrolled in the cardiopulmonary substudy with evaluable baseline echocardiogram scans per the central laboratory) and with both baseline and at least one post-baseline LVEF measurement within 24 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 40 | 48
percentage of participants | 2.6 | 0.0

7. Secondary Outcome: Change From Baseline in Right Ventricular Fractional Area Change (FAC)
Description: Right ventricular function was assessed by measuring fractional area change (FAC) on echocardiogram.
Time Frame: Baseline and Weeks 12, 24 and 36 and at end of treatment (median duration of treatment was 27 weeks in the bortezomib group and 40 weeks in the carfilzomib treatment group).
Population: Cardiopulmonary Safety Evaluable subgroup with available FAC data at baseline; "n" indicates participants whose results were available at both the baseline and the specified post-baseline visit.
Measure: Mean (Standard Deviation); unit: percent fractional area change
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 52 | 55
percent fractional area change
  Week 12 (n=40, 40) | -0.7 (5.00) | -1.1 (5.36)
  Week 24 (n=26, 31) | 0.7 (6.10) | -1.0 (5.03)
  Week 36 (n=15, 18) | -0.5 (7.27) | -0.5 (6.38)
  End of Treatment (n=23, 18) | 0.4 (4.73) | -1.9 (5.47)

8. Secondary Outcome: Change From Baseline in Pulmonary Artery Systolic Pressure (PASP)
Description: Pulmonary artery pressure was measured using transthoracic echocardiogram.
Time Frame: as for outcome 7
Population: Cardiopulmonary Safety Evaluable subgroup with available PASP data at baseline; "n" indicates participants whose results were available at both the baseline and the specified post-baseline visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bortezomib + DEX | Carfilzomib + DEX
Number analyzed (Participants) | 52 | 45
mmHg
  Week 12 (n=34, 30) | 0.3 (11.72) | 2.8 (11.44)
  Week 24 (n=22, 20) | 1.7 (8.47) | 3.4 (13.63)
  Week 36 (n=12, 14) | 4.0 (7.24) | 2.6 (13.55)
  End of Treatment (n=21, 14) | 3.4 (8.14) | 0.9 (11.40)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug as of the data cut-off date of 03 January 2017; median duration of treatment was 27 weeks in the bortezomib group and 48 weeks in the carfilzomib treatment group.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Bortezomib | Carfilzomib
Serious Adverse Events (participants affected / at risk) | 182/456 | 272/463
Other Adverse Events (participants affected / at risk) | 435/456 | 446/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=456) | Carfilzomib (N=463)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 3
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
PLASMACYTOSIS (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 4
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 0 | 2
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 2
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 3
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 6
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
BIFASCICULAR BLOCK (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 2
CARDIAC FAILURE (Cardiac disorders) | 3 | 9
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CARDIAC HYPERTROPHY (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 2
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 5
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
PLEUROPERICARDITIS (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 2
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 | 0
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 0
RETINAL TEAR (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 11 | 5
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
ILEUS PARALYTIC (Gastrointestinal disorders) | 3 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL POLYP HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 2
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 1 | 1
VOMITING (Gastrointestinal disorders) | 2 | 5
ASTHENIA (General disorders) | 1 | 0
CARDIAC DEATH (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 4 | 3
DEATH (General disorders) | 0 | 1
DEVICE OCCLUSION (General disorders) | 1 | 0
DISEASE PROGRESSION (General disorders) | 6 | 8
FATIGUE (General disorders) | 1 | 3
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 4
GENERALISED OEDEMA (General disorders) | 1 | 0
HYPERPYREXIA (General disorders) | 1 | 0
HYPERTHERMIA (General disorders) | 0 | 1
MALAISE (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 3 | 19
SUDDEN DEATH (General disorders) | 1 | 3
THROMBOSIS IN DEVICE (General disorders) | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 2
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1
LIVER DISORDER (Hepatobiliary disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 | 1
ABDOMINAL INFECTION (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
BACTERIAL DIARRHOEA (Infections and infestations) | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 2 | 1
BREAST ABSCESS (Infections and infestations) | 1 | 0
BRONCHIOLITIS (Infections and infestations) | 0 | 2
BRONCHITIS (Infections and infestations) | 2 | 8
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 7
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
BURSITIS INFECTIVE (Infections and infestations) | 1 | 1
CATHETER SITE INFECTION (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 3
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE SEPSIS (Infections and infestations) | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 2
DIVERTICULITIS (Infections and infestations) | 0 | 3
ENCEPHALITIC INFECTION (Infections and infestations) | 0 | 1
ENCEPHALITIS HERPES (Infections and infestations) | 0 | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
FEBRILE INFECTION (Infections and infestations) | 0 | 2
GASTROENTERITIS (Infections and infestations) | 4 | 5
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1
H1N1 INFLUENZA (Infections and infestations) | 0 | 1
HAEMOPHILUS SEPSIS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 4
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 1
INFLUENZA (Infections and infestations) | 1 | 3
LISTERIOSIS (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 1 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 7
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 3 | 5
NECROTISING ULCERATIVE PERIODONTITIS (Infections and infestations) | 0 | 1
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 1
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 | 2
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMOCOCCAL INFECTION (Infections and infestations) | 0 | 1
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 42 | 39
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1
PNEUMONIA MORAXELLA (Infections and infestations) | 1 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 | 1
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 | 0
PULMONARY SEPSIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 2 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 10
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 2
SEPSIS (Infections and infestations) | 4 | 7
SEPTIC SHOCK (Infections and infestations) | 3 | 4
SINUSITIS (Infections and infestations) | 0 | 1
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 7
URINARY TRACT INFECTION (Infections and infestations) | 4 | 6
UROSEPSIS (Infections and infestations) | 3 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 3
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 3
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0
OPEN WOUND (Injury, poisoning and procedural complications) | 1 | 0
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD CORTISOL DECREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 2
INFLUENZA B VIRUS TEST POSITIVE (Investigations) | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 3 | 2
TROPONIN T INCREASED (Investigations) | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 2
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 5 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 6
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 4
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 2
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MENINGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
OESOPHAGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
PLEURAL MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ACQUIRED EPILEPTIC APHASIA (Nervous system disorders) | 0 | 1
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 4
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 2
HYPERCAPNIC COMA (Nervous system disorders) | 0 | 1
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 3
LETHARGY (Nervous system disorders) | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
NEURALGIA (Nervous system disorders) | 1 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 1
PARAPARESIS (Nervous system disorders) | 1 | 0
PARAPLEGIA (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 | 2
RADICULITIS BRACHIAL (Nervous system disorders) | 0 | 1
RADICULOPATHY (Nervous system disorders) | 0 | 1
SCIATICA (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 2 | 4
SYNCOPE (Nervous system disorders) | 4 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 4 | 4
DEPRESSION (Psychiatric disorders) | 1 | 1
DYSTHYMIC DISORDER (Psychiatric disorders) | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1
ALBUMINURIA (Renal and urinary disorders) | 0 | 1
ANURIA (Renal and urinary disorders) | 0 | 1
NEPHROPATHY (Renal and urinary disorders) | 1 | 1
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 5
RENAL FAILURE ACUTE (Renal and urinary disorders) | 7 | 11
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 18
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 10
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 4
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1
COLOSTOMY CLOSURE (Surgical and medical procedures) | 0 | 1
HAEMORRHOID OPERATION (Surgical and medical procedures) | 0 | 1
REMOVAL OF INTERNAL FIXATION (Surgical and medical procedures) | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 0 | 1
AORTIC EMBOLUS (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 5
HAEMATOMA (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 3
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 4 | 1
MALIGNANT HYPERTENSION (Vascular disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 4 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 2
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=456) | Carfilzomib (N=463)
ANAEMIA (Blood and lymphatic system disorders) | 129 | 196
LYMPHOPENIA (Blood and lymphatic system disorders) | 25 | 31
NEUTROPENIA (Blood and lymphatic system disorders) | 26 | 27
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 83 | 100
CATARACT (Eye disorders) | 17 | 32
CONJUNCTIVITIS (Eye disorders) | 36 | 22
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 26 | 20
ABDOMINAL PAIN (Gastrointestinal disorders) | 38 | 32
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 35 | 24
CONSTIPATION (Gastrointestinal disorders) | 126 | 75
DIARRHOEA (Gastrointestinal disorders) | 184 | 167
DYSPEPSIA (Gastrointestinal disorders) | 25 | 35
NAUSEA (Gastrointestinal disorders) | 89 | 108
VOMITING (Gastrointestinal disorders) | 44 | 75
ASTHENIA (General disorders) | 78 | 107
CHEST PAIN (General disorders) | 19 | 42
CHILLS (General disorders) | 12 | 26
FATIGUE (General disorders) | 140 | 149
INFLUENZA LIKE ILLNESS (General disorders) | 10 | 24
MALAISE (General disorders) | 8 | 24
OEDEMA PERIPHERAL (General disorders) | 87 | 116
PYREXIA (General disorders) | 68 | 144
BRONCHITIS (Infections and infestations) | 46 | 103
NASOPHARYNGITIS (Infections and infestations) | 61 | 81
PNEUMONIA (Infections and infestations) | 18 | 24
RESPIRATORY TRACT INFECTION (Infections and infestations) | 29 | 47
RHINITIS (Infections and infestations) | 10 | 29
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 80 | 116
URINARY TRACT INFECTION (Infections and infestations) | 28 | 34
CONTUSION (Injury, poisoning and procedural complications) | 25 | 19
FALL (Injury, poisoning and procedural complications) | 23 | 18
BLOOD CREATININE INCREASED (Investigations) | 28 | 52
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 18 | 29
LYMPHOCYTE COUNT DECREASED (Investigations) | 18 | 42
PLATELET COUNT DECREASED (Investigations) | 41 | 57
DECREASED APPETITE (Metabolism and nutrition disorders) | 61 | 50
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 42 | 53
HYPERURICAEMIA (Metabolism and nutrition disorders) | 8 | 31
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 19 | 27
HYPOKALAEMIA (Metabolism and nutrition disorders) | 51 | 60
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 28 | 32
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 51 | 60
BACK PAIN (Musculoskeletal and connective tissue disorders) | 81 | 105
BONE PAIN (Musculoskeletal and connective tissue disorders) | 40 | 55
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 28 | 92
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 47 | 44
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 20 | 39
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 23 | 24
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 28
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 50 | 55
DIZZINESS (Nervous system disorders) | 69 | 42
DYSGEUSIA (Nervous system disorders) | 27 | 16
HEADACHE (Nervous system disorders) | 49 | 95
HYPOAESTHESIA (Nervous system disorders) | 14 | 24
NEURALGIA (Nervous system disorders) | 72 | 11
NEUROPATHY PERIPHERAL (Nervous system disorders) | 130 | 49
PARAESTHESIA (Nervous system disorders) | 76 | 43
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 70 | 29
POLYNEUROPATHY (Nervous system disorders) | 26 | 6
TREMOR (Nervous system disorders) | 23 | 10
ANXIETY (Psychiatric disorders) | 33 | 19
INSOMNIA (Psychiatric disorders) | 122 | 125
COUGH (Respiratory, thoracic and mediastinal disorders) | 72 | 128
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 62 | 144
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 14 | 24
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 19 | 28
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 15 | 27
PRURITUS (Skin and subcutaneous tissue disorders) | 29 | 34
RASH (Skin and subcutaneous tissue disorders) | 35 | 41
FLUSHING (Vascular disorders) | 7 | 24
HYPERTENSION (Vascular disorders) | 45 | 148
HYPOTENSION (Vascular disorders) | 37 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.